CLINICAL TRIAL: NCT04030117
Title: Clinical and Radiographic Assessment of Bioactive Restorative Material Versus Polyacid Modified Composite Resin in Treatment of Class II Restorations in Primary Molars: A Pilot Study
Brief Title: Class II Restoration Using Bioactive Restorative Material vs Polyacid Modified Composite Resin in Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Mohsen Ahmed Moustafa, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19121987
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Class II Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTIVA Test arm (Experimental): Treatment of decay in Class II second primary molars using ACTIVA restorative material.
  Interventions: Procedure: ACTIVA Bioactive restoration
- Compomer Comparator arm (Active Comparator): Treatment of decay in Class II second primary molars using compomer restorative material.
  Interventions: Procedure: Compomer restoration

INTERVENTIONS:
Procedure: ACTIVA Bioactive restoration — Removal of Class II decay in second primary molars and placement of ACTIVA restoration.
  Other Names: ACTIVA Bioactive Class II restoration
  Arms: ACTIVA Test arm
Procedure: Compomer restoration — Removal of Class II decay in second primary molars and placement of Compomer restoration.
  Other Names: Compomer Class II restoration
  Arms: Compomer Comparator arm

SUMMARY:
Successful restoration of cavities in primary molars can be considered challenging. It is different from restoring cavities in permanent molars because factors such as the level of co-operation of the child and the handling properties and setting time of the restorative material will have some influence on the success rate of the restoration. The ideal requirements that a filling material should possess include that it bears the occlusal force, withstands the acidic and bacterial attack, survives in the oral environment in addition to being biocompatible with the oral tissues.

In an attempt to achieve this idealism, a new class of restorative materials known as "bioactive materials" has been developed. The concept of bioactive materials was introduced in 1969 and later defined as "one that elicits a specific biological response at the interface of the material which results in the formation of a bond between tissues and the material." An example of bioactive materials is ACTIVA™ BioACTIVE (Pulpdent, USA). These materials are ionic composite resins which combine the biocompatibility, chemical bond and the ability to release fluoride of glass ionomers with the mechanical properties, esthetic and durability of composite resins.

Compomer is widely accepted as a standard restorative material for primary dentition for Class I and II cavities. Its range of success rate in Class II restorations in primary molars is 78-96%. Many randomized clinical trials have reported comparable clinical performance to composite resin with respect to color matching, marginal discoloration, anatomical form, marginal integrity and secondary caries. In comparison to glass ionomer and Resin Modified Glass Ionomer, compomers tend to have better physical properties in the primary dentition. However, their cariostatic properties didn't differ significantly from those materials.

DETAILED DESCRIPTION:
1. Hypothesis:

   The null hypothesis is that there is no difference between using ACTIVA and Dyract® in children to restore Class II cavities in carious vital primary second molars.
2. Trial design:

   * A pilot study, parallel group, two arm.
   * Allocation ratio is 1:1.
3. Method

Intervention:

A) Diagnosis:

* Diagnostic chart will be filled with personal, medical and dental history.
* The intra-oral examination will be made using gloves, mask, gauze and dental mirror.
* A pre-operative radiograph (bitewing) will be taken for diagnosis. b) The intervention in this pilot study will be (ACTIVA™ BioACTIVE, Pulpdent, USA) - Gp1 while the comparator will be (Dyract® DENTSPLY, Germany)- Gp2.

Three follow up visits for restoration at:

T1 (3 months), T2 (6 months) and T3 (12 months).

Same procedure in both groups will be followed:

1. The tooth will be anesthetized using local anesthesia, and isolated using rubber dam.
2. Caries will be removed.
3. A proximal box is prepared.
4. A metal matrix band is fixed around the tooth and a wedge is placed interdentally.
5. The restorative material chosen according to the randomization is placed in the cavity according to the manufacturer's instructions.
6. A post-operative digital bitewing radiograph will be taken immediately after the treatment as a base line reference and to check for voids or any defect in the restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Children with Class II cavities in vital primary second molars.
2. Proximal enamel/dentin caries limited to outer half of dentin.
3. Age ranging from 4-8 years.
4. Good general health.

Exclusion Criteria:

1. Spontaneous pain related to carious molars.
2. Abscess or fistula on examination or during history taking.
3. Tooth mobility.
4. Radiographic evidence of root resorption or close shedding time.
5. Lack of patient co-operation.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative sensitivity | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration, Bravo (B) = acceptable clinical situation, and Charlie (C) = clinically unacceptable restorations (failure).

SECONDARY OUTCOMES:
Color match | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration, Bravo (B) = acceptable clinical situation, and Charlie (C) = clinically unacceptable restorations (failure).
Marginal discoloration | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration, Bravo (B) = acceptable clinical situation, and Charlie (C) = clinically unacceptable restorations (failure).
Marginal adaptation (integrity) | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration, Bravo (B) = acceptable clinical situation, and Charlie (C) = clinically unacceptable restorations (failure).
Surface texture | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration, Bravo (B) = acceptable clinical situation, and Charlie (C) = clinically unacceptable restorations (failure).
Anatomic form | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration, Bravo (B) = acceptable clinical situation, and Charlie (C) = clinically unacceptable restorations (failure).
Gross/restoration fracture | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration, Bravo (B) = acceptable clinical situation, and Charlie (C) = clinically unacceptable restorations (failure).
Tooth fracture | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration, Bravo (B) = acceptable clinical situation, and Charlie (C) = clinically unacceptable restorations (failure).
Secondary caries | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration and (C) = clinically unacceptable restorations (failure).
Pulpal affection | 12 months
  Using modified United States health service (USPHS)/ Ryge criteria. Scores: Alpha (A) = Ideal clinical restoration and (C) = clinically unacceptable restorations (failure).

OTHER OUTCOMES:
Secondary/recurrent caries | 12 months
  Using standardized bite-wing radiograph to check presence or absence of secondary caries.

CONTACTS AND LOCATIONS:
Overall Officials: Cairo University, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
After thesis defense the study will be published internationally to be available for the public.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within one year and a half
Access Criteria: Not yet